CLINICAL TRIAL: NCT02619734
Title: Efficacy and Safety of Autologous Bone Marrow Stem Cells Infusion for Treatment of Chronic Leg Ulcer in Sickle Cell Disease Patients
Brief Title: Autologous Bone Marrow Stem Cells for Chronic Leg Ulcer Treatment in Sickle Cell Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Bahia (Other)
Collaborators: Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Vitor Fortuna, PhD, Federal University of Bahia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11738
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Leg Ulcer; Sickle Cell Disease
Keywords: Cell Therapy; Sickle cell disease; Autologous implantation; Mesenchymal stromal cell; Edothelial Progenitor cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Conventional treatment established by the good clinical practice Patients received standard local care dressing method (compresses) to heal leg ulcers
- Stem Cell Injection (Experimental): Intramuscular implantation of Autologous bone marrow-derived mononuclear cells
  Interventions: Biological: Infusion of Autologous Bone Marrow Mononuclear Cells

INTERVENTIONS:
Biological: Infusion of Autologous Bone Marrow Mononuclear Cells — Autologous bone marrow-derived mononuclear cells will be administered by intramuscular injection into and around the leg ulcer. The number of injected cells will be from 5x108 to 1x109 total number of cells on Study Day 1.
  Arms: Stem Cell Injection

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of autologous bone marrow stem cell implantation for the treatment of leg ulcer in adult patients with sickle cell disease.

DETAILED DESCRIPTION:
Implantation of bone marrow mononuclear cells, including endothelial progenitor cells and mesenchymal stromal cells, into leg ulcers has been shown to improve wound healing.

In the present study the safety and efficacy of autologous bone marrow mononuclear cells implantation will be investigated in patients with chronic leg ulcers. Forty cases will be enrolled. Improvement in the pain, rate and extent of leg ulcer wound healing as measured by change in wound surface area will be evaluated until one year.

ELIGIBILITY:
Inclusion Criteria:

* Stable sickle cell disease patients
* Patient hospitalized into the dermatology unit
* Patient with an evolutive leg ulcer since more than 1 year
* No infection at the time of surgery
* Patient competent to give informed consent

Exclusion Criteria:

* Patients with a history of corticosteroids or on active therapy
* infection at the limb affected by ulcer
* Recurrent painful crises,
* Immunosuppressive drug therapy,
* Pregnancy,
* Presence of neoplastic disease or any other clinical concurrent condition other than sickle cell disease that predisposed them to the development of leg ulcer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Safety of Treatment - Determined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis measures, and reported adverse events | 6 months
  Determined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis measures, and reported adverse events
Change in Leg Ulcer | 6 months to one year
  Rate and extent of leg ulcer wound healing as measured by change in wound surface area Ulcer diameter will be recorded

SECONDARY OUTCOMES:
Numeric pain intensity scale (0-10) | 6 months to one year
  Change in Sickle Cell Disease leg ulcer wound pain scores as measured by a 10-point scale (analogic visual scale) and relative to non-wound site pain scores
Ulcer Healing | 6 months to one year
  Defined as a Decrease in Ulcer Area by at Least 25% of the Initial Area Ulcer diameter will be recorded
Quality of Life | 6 months to one year
  Change in quality of life as well as other indicators of patient comfort and well-being

CONTACTS AND LOCATIONS:
Overall Officials: José Valber Meneses, MD, Study Chair — Federal University of Bahia; Gildasio Daltro, MD, Study Director — Federal University of Bahia; Vitor A Fortuna, PhD, Principal Investigator — Federal University of Bahia

REFERENCES:
- [Background] Daltro GC, Fortuna V, de Souza ES, Salles MM, Carreira AC, Meyer R, Freire SM, Borojevic R. Efficacy of autologous stem cell-based therapy for osteonecrosis of the femoral head in sickle cell disease: a five-year follow-up study. Stem Cell Res Ther. 2015 May 29;6(1):110. doi: 10.1186/s13287-015-0105-2. PMID 26021713